CLINICAL TRIAL: NCT00313729
Title: A Phase II Study of Temozolomide (TEMODAR) in the Treatment of Adult Patients With Supratentorial Low Grade Glioma
Brief Title: Temozolomide in Treating Patients With Low-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Susan Chang, MD, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000448883; 99102 (Other: UCSF Cancer Center Protocol Number); BTRC-9902; H7858-16278-07 (Other: UCSF IRB); NCT00187642 (obsolete NCT alias)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-01

CONDITIONS: CNS Tumor, Adult
Keywords: adult oligodendroglioma; adult mixed glioma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Glioma; Astrocytoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental): Temozolomide
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — Chemotherapy
  Other Names: Temodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well temozolomide works in treating patients with supratentorial low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of temozolomide, defined as response rate (complete and partial response), in patients with supratentorial mixed low-grade glioma.

Secondary

* Assess the safety profile of temozolomide in patients with supratentorial low-grade glioma.
* Assess the time to tumor progression in patients treated with temozolomide.

OUTLINE: Patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven supratentorial low-grade (grade II) glioma of any of the following histologic subtypes:

  * Oligodendroglioma
  * Astrocytoma
  * Oligoastrocytoma
* Has undergone surgical resection or biopsy within 35 days after diagnosis of low-grade glioma

  * Study treatment must begin between 14 days and 4 months after surgical resection or biopsy
* Evaluable disease by gadolinium-MRI

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine < 1.5 times upper limit of normal (ULN)
* BUN < 1.5 times ULN
* Bilirubin < 1.5 times ULN
* SGOT < 2.5 times ULN
* Alkaline phosphatase < 2 times ULN
* Life expectancy > 12 weeks
* No nonmalignant systemic disease resulting in the patient being a poor medical risk
* No acute infection requiring intravenous antibiotics
* No frequent vomiting or medical condition that would interfere with oral medication intake (e.g., partial bowel obstruction)
* No other concurrent malignancies except surgically cured carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin

  * Prior malignancies must be in remission for ≥ 5 years
* No known HIV positivity
* No AIDS-related illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy, interstitial brachytherapy, or radiosurgery for low-grade glioma
* No prior biological therapy or chemotherapy for low-grade glioma
* No other concurrent chemotherapy
* No concurrent radiotherapy or biological therapy
* No concurrent prophylactic growth factors
* No concurrent epoetin alfa
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1999-05; Primary Completion 2014-09-25 (Actual); Study Completion 2017-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Chang, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Study of Temozolomide for LGG Patients: Oral temozolomide at 200mg/m2 per day x5 days every 28 days for up to 12 cycles
Period: Overall Study
Arm/Group | Single Arm Study of Temozolomide for LGG Patients
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Temozolomide: Single Arm Trial with single dose schedule of Temozolomide chemotherapy
Arm/Group | Temozolomide
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 119
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial Response)
Description: Assessment of treatment response was determined by MRI in conjunction with neurological examination and steroid requirement assessment derived from Macdonald's criteria. Complete response was defined as complete disappearance of lesion on consecutive MRI scans with stable or improved neuro exam and steroids. Partial response was defined as a 50% reduction in lesion size or that tumor burden was "definitely better" than prior scan with stable or improved neuro exam and steroids.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 120
Participants | 7

2. Secondary Outcome: Time to Tumor Progression
Description: Progressive disease was defined as definite enlargement of any existing lesion or any new lesion based on modified Macdonald's criteria.
Time Frame: time from registration until date of the first documented progression, an average of 1 year
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Temozolomide
Number analyzed (Participants) | 120
years | 3.8 [3.0 to 5.0]

3. Secondary Outcome: Safety Profile
Description: Number of participants with treatment related grade 2-4 adverse events as defined by CTCAE 3.0
Time Frame: Time from registration up to 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 120
Participants | 12

ADVERSE EVENTS:
Arm/Group | Temozolomide
Serious Adverse Events (participants affected / at risk) | 17/120
Other Adverse Events (participants affected / at risk) | 31/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=120)
Neutrophils/granulocytes (ANC) (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (platelets) (Blood and lymphatic system disorders) | 1 (1) — Grade 4
Infection with unknown ANC (Infections and infestations) | 1 (1)
seizure (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1) — Grade III
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade III
Death (Nervous system disorders) | 1 (1) — Death within 30 days of study drug - unlikely related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=120)
Fatigue (Metabolism and nutrition disorders) | 9 (18) — Constitutional Symptoms: Fatigue (asthenia, lethargy, malaise)
Nausea (Gastrointestinal disorders) | 11 (17)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5 (6)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Seizures (Nervous system disorders) | 7 (8) — Neurology
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (5)
Tremor (Nervous system disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 5 (11)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (22)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 (19)
Platelets (Blood and lymphatic system disorders) | 5 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Insomnia (Nervous system disorders) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Memory loss (Nervous system disorders) | 1 (1) — Memory impairment
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (2)
GGT (γ-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Neuropathy: cranial (Nervous system disorders) | 1 (1)
Pain - Other (General disorders) | 5 (7)
Hemoglobin (Blood and lymphatic system disorders) | 2 (3)
Rash: dermatitis associated with high-dose chemotherapy or BMT studies (Skin and subcutaneous tissue disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6) — Glucose, serum-high (hyperglycemia)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Personality/behavioral (Nervous system disorders) | 1 (1)
Mood alteration - depression (Nervous system disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 (1) — Mucositis/stomatitis
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound-infectious (Infections and infestations) | 1 (1) — Infection - Select
diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (1) — diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No